CLINICAL TRIAL: NCT06185842
Title: The Effectiveness of a Comprehensive Lung Health Promotion Program Based on the 5A Self-management Support Model for the Elderly in Nursing Home: A Randomized Controlled Trial.
Brief Title: The Effectiveness of a Lung Health Promotion Program Based on the 5A Self Management Support Model.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, NURSEZA AKGÖZ, Research Assistant, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SelcukU-nursing-NA-01
Record Dates: First submitted 2023-12-16; First posted 2023-12-29 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2023-11

CONDITIONS: Pulmonary Disease
MeSH Terms: conditions — Lung Diseases | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): breathing exercise, walking exercise and vaccination counseling
  Interventions: Behavioral: breathing exercise, walking exercise and vaccination counseling
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: breathing exercise, walking exercise and vaccination counseling — Participants will perform diaphragmatic breathing exercises and pursed lip breathing exercises two days a week for eight weeks.
  Participants will be asked to walk for 20-30 minutes every day for eight weeks. Monitoring will be done weekly.
  Participants will be counseled about infectious diseases, modes of transmission and the importance of vaccination, and will be advised to receive influenza and pneumococcal vaccines recommended for this age group.
  The 5A model guide will be used regarding behavioral change towards physical activity and vaccination.
  Arms: Intervention group

SUMMARY:
This research will be conducted to examine the effect of the lung health promotion program based on the 5A self-management support model on some physiological parameters, Physical Activity Scale in the Elderly score, sleep quality, health status perception and vaccination status of adults aged 65 and over.

The research will be carried out as a randomized controlled study with a parallel design.

We estimate that the respiratory functions of the elderly will improve, their physical activity levels will increase, immunization against common infectious diseases will increase and people's health perceptions will improve. with the lung health promotion program based on the 5A self-management support model.

DETAILED DESCRIPTION:
The population of the research consisted of 312 individuals aged 60 and over living in an elderly care and rehabilitation center.

In the sample calculation of the research, taking into account the GPower 3.1.9.7 program and the results of similar studies in the literature, it was calculated that it would be sufficient to include a total of 42 individuals, 21 elderly individuals in each group, with a margin of error of 0.05 and a test power of 80%.

Considering that there may be losses during the process in such studies, 5% of the sample number (2.1~2 people) was added to the study. The study was planned to include 22 elderly individuals in the intervention group and 22 elderly individuals in the control group.

A program to improve lung health will be applied to the elderly in the experimental group.

Within the scope of the research, participants; They will do diaphragmatic breathing exercises and pursed lip breathing exercises 2 days a week for 8 weeks.

Participants will be asked to walk for 20-30 minutes every day for eight weeks. Monitoring will be done weekly.

Participants will be counseled about infectious diseases, modes of transmission and the importance of vaccination, and will be advised to receive influenza and pneumococcal vaccines recommended for this age group.

The 5A model guide will be used regarding behavioral change towards physical activity and vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Being 60 years or older
* Being literate / Being able to read and write Turkish
* Scoring 24 or above on the Standardize Mini Mental Test Examination
* No bilateral vision or bilateral hearing problems
* Not having an acute or chronic systemic disease that would prevent breathing exercise (pulmonary hypertension, angina pectoris, recent myocardial infarction, aortic stenosis, congestive heart failure, heart valve disease, abdominal aortic aneurysm, unstable diabetes, hypoxemia that cannot be corrected by oxygen supplementation due to heavy exercise, severe peripheral vascular disease, recent deep vein thrombosis etc.)
* Having no musculoskeletal system problems that prevent walking (arthritis, musculoskeletal injuries etc.)
* Not having had a recent surgical intervention (cataract surgery, ear, brain, spinal cord surgery, diaphragmatic rupture, hiatus or abdominal hernia repair surgery etc.)
* Not having severe liver disease and active substance addiction
* Not having advanced dementia, cognitive and psychological disorders, psychiatric diseases and serious neurological diseases.

Exclusion Criteria:

* Having an acute problem or complication related to existing chronic diseases
* Withdrawing from the research voluntarily. However, the data of this group of elderly people will be analyzed with intention to treat (ITT) analysis.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
6-minute walk distance | 8 weeks
  The six-minute walk test (6MWT) is an exercise test used to evaluate walking endurance and aerobic capacity. This test measures the distance the patient can walk quickly on a flat, hard surface in a 6-minute period.
  It is reported that the distance walked for six minutes varies between 400-700m in normal individuals.
  The distance the person is expected to walk during the test is calculated based on age, gender, height and body mass index. It is accepted that the distance recorded in the test provides information about the person's exercise capacity during daily living activities.
forced vital capacity (FVC) | 8 weeks
  FVC-Forced vital capacity; the total volume of air that can be exhaled during a maximal forced expiration effort.
forced expiratory volume in one second (FEV1) | 8 weeks
  FEV1-Forced expiratory volume in one second; the volume of air exhaled in the first second under force after a maximal inhalation.
FEV1/FVC ratio | 8 weeks
  FEV1/ FVC ratio-The percentage of the FVC expired in one second.
Physical Activity Scale for the Elderly (PASE) | 8 weeks
  The PASE was developed for the purpose of evaluating the components of physical activities involving leisure time, work-related activities, and the household.
  The PASE is a self-reported questionnaire that consists of 12 questions regarding the frequency and duration of leisure time activity, household activity, and work-related activity during the previous 7-day period.
  The questions are scored differently. Participation in leisure time and strengthening activities are scored as never, seldom (1 or 2 days per week), sometimes (3 or 4 days per week), and often (5-7 days per week). Duration of these activities is scored as less than 1 h, 1-2 h, 2-4 h, and more than 4 h.
  The overall PASE score ranges from 0 to 400 or more and high scores show better physical activity levels.
health status perception | 8 weeks
  To determine their perception of health status, participants are asked to evaluate their general health status over the past 15 days using a visual analog scale.
  Accordingly, the participant marks an integer score from 0 to 10 according to the following five categories: 0 = terrible, 1- 3 = poor, 4-6 = fair, 7-9 = good, and 10 = excellent.
sleep quality | 8 weeks
  The single-item sleep quality scale (SQS) is a practical measurement tool that can effectively measure sleep quality in the clinical setting.
  A visual analog scale is used to rate the individual's overall sleep quality over the past seven days.
  In this way, the participant marks an integer score from 0 to 10 according to the following five categories: 0 = terrible, 1- 3 = poor, 4-6 = fair, 7-9 = good, and 10 = excellent.
  When rating their sleep quality, participants are asked to consider the following key components of sleep quality: how many hours they slept, how easily they fell asleep, how often they woke up during the night (other than to go to the toilet), how often they woke up early in the morning, and how restful their sleep was.

CONTACTS AND LOCATIONS:
Overall Officials: NURSEZA AKGÖZ, PhD, Principal Investigator — Selcuk University
Locations (1):
- Dr. İsmail Işık Huzurevi Yaşlı Bakım ve Rehabilitasyon Merkezi, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No